CLINICAL TRIAL: NCT03129594
Title: Prognostic Value of Plasma Glucagon-like Peptide-1 Levels in Acute Myocardial Infarction
Brief Title: Plasma Glucagon-like Peptide-1 Levels and Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Jing Wei, Doctor, Chinese PLA General Hospital
Other Study IDs: GLP1AMI
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Coronary Angiography; Glucagon-like Peptide-1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: plasma glucagon-like peptide-1 levels — The plasma GLP-1 levels was determined by enzymatic assays.

SUMMARY:
GLP-1(9-36) amide and (9-37), which was previously thought to be the inactive metabolite of GLP-1, also exerts cardioprotective effects. Direct administration of GLP-1(9-36) during reperfusion reduced ischaemic damage in isolated hearts and increased cGMP release, vasodilatation and coronary flow in AMI mouse model, one may speculate that total GLP-1 level may associate with adverse cardiovascular events in AMI patients, the hypothesis is therefore tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients of acute AMI come to our department,absent of cardiogenic shock, and survival for at least 24 h after PCI treatment.

Exclusion Criteria:

* patients with cancer, and patients who were taking a DPP4 inhibitor or a glucagon-like peptide-1 (GLP-1) analogue

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A single center study on PCI-treated myocardial infarction patients
Sampling Method: Non-Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | The median follow-up was 29 months
cardiovascular mortality | The median follow-up was 29 months

SECONDARY OUTCOMES:
non-cardiovascular mortality | The median follow-up was 29 months
Myocardial infarction | The median follow-up was 29 months
heart failure readmission | The median follow-up was 29 months
  readmission to any hospital due to diagnosed heart failure
Stroke | The median follow-up was 29 months
  defined using the World Health Organization criteria
repeated revascularization | The median follow-up was 29 months
  defined as repeated PCI or bypass grafting of not only infarct related artery